CLINICAL TRIAL: NCT00171457
Title: The Effects of Tegaserod on Mechanical Sensitivity of the Esophagus and Stomach in Patients With Heartburn and Dyspepsia.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CHTF919DUS45
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2007-10-10 (Estimated); Status verified 2007-10

CONDITIONS: Heartburn; Dyspepsia
Keywords: functional heartburn; dyspepsia; male; female; visceral sensitivity
MeSH Terms: conditions — Heartburn; Dyspepsia | interventions — tegaserod

INTERVENTIONS:
Drug: Tegaserod

SUMMARY:
Investigate the role of tegaserod in modulating gastric sensitivity to mechanical distention of the stomach

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects at least 18 years of age.
* Subjects willing to undergo multiple nasogastric intubations.
* Patients with functional heartburn will need to meet ROME II criteria.
* Patients with symptoms consistent with dyspepsia (epigastric pain/discomfort characterized by bloating, postprandial fullness and early satiety)

Exclusion Criteria:

* Subjects with clinically significant diarrhea or a diagnosis of diarrhea-predominant IBS.
* Subjects with a diagnosis of IBD, Barrett's esophagus, esophageal stricture or ring, or previous or current history of ulcer disease.
* Subjects with Diffuse Esophageal Spasm or Achalasia.

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 24
Dates: Start 2005-04; Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
To determine if tegaserod 6 mg b.i.d modulates gastric sensitivity to mechanical distention of the stomach

SECONDARY OUTCOMES:
1) Comparing effects at end of treatment compared to baseline:
To verify that tegaserod modulates esophageal sensitivity to esophageal distention
To determine if tegaserod improves individual dyspeptic symptoms of epigastric pain/discomfort
To determine if tegaserod improves heartburn and/or regurgitation
To determine if tegaserod is preferred by patients with functional heartburn & accompanying dyspepsia & gastric mechanical sensitivity over placebo
Safety assessment
To determine if there is a correlation between esophageal & gastric mechanosensitivity thresholds in this patient group, and to determine if tegaserod alters this relationshi

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Director — Novartis
Locations (1):
- Oklahoma Foundation for Digestive Research, Oklahoma City, Oklahoma, United States

REFERENCES:
- [Derived] Miner PB Jr, Rodriguez-Stanley S, Proskin HM, Kianifard F, Bottoli I. Tegaserod in patients with mechanical sensitivity and overlapping symptoms of functional heartburn and functional dyspepsia. Curr Med Res Opin. 2008 Aug;24(8):2159-72. doi: 10.1185/03007990802222832. Epub 2008 Jun 17. PMID 18561877